CLINICAL TRIAL: NCT02155361
Title: Evaluation of Topical Citrullus Colocynthis Fruit Oil Efficacy in Treatment of Painful Peripheral Diabetic Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Dr. Mesbah Shams, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-9377-7007
Record Dates: First submitted 2014-05-31; First posted 2014-06-04 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetes mellitus; Diabetes complications; Pain
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Diabetes Complications; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Citrullus colocynthis fruit oil (Active Comparator): Topical Citrullus colocynthis fruit oil (1%) 1 cc twice daily
  Interventions: Drug: Topical Citrullus colocynthis fruit oil (1%)
- Placebo (Vehicle) (Placebo Comparator): Topical vehicle oil 1 cc twice daily
  Interventions: Drug: Topical vehicle oil

INTERVENTIONS:
Drug: Topical Citrullus colocynthis fruit oil (1%)
  Arms: Topical Citrullus colocynthis fruit oil
Drug: Topical vehicle oil
  Arms: Placebo (Vehicle)

SUMMARY:
This study is designed to evaluate the topical Citrullus colocynthis fruit oil efficacy in treatment of painful peripheral diabetic neuropathy (PDN) in a randomized double blind placebo-controlled clinical trial design. This study includes 60 patients from SUMS endocrinology and diabetes clinic. Patients with painful conditions other than PDN such as radiculopathies will be excluded. After giving the Informed consent the patients will be underwent NCS (Nerve Conduction Study) for confirming the diagnosis before recruitment. They will be followed for 12 weeks and after 12 weeks the outcome measures including Neuropathic Pain Scale (NPS), WHOQOL-BREF (World Health Organisation Quality of Life Brief) questionnaire and electrodiagnostic criteria will be evaluated.

ELIGIBILITY:
Inclusion criteria:

* Controlled type 1 or 2 diabetes mellitus
* Painful Peripheral diabetic neuropathy for more than 3 months
* Age more than 18 years old
* Patients consent on enrolling study and admitting study protocol

Exclusion criteria:

* Other causes of pain in lower extremities like lumbar disk herniation
* Ulcerative lesions in lower extremities
* Dermatitis
* Pregnancy
* Lactation
* Citrullus colocynthis allergy
* Unstable cardiac, neurological or renal disease
* Diagnosed other types of neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Neuropathic Pain Scale (NPS) | 12 weeks

SECONDARY OUTCOMES:
WHOQOL-BREF Score | 12 weeks
Number of Participants with Adverse Events | 12 weeks
Nerve Conduction Velocity (NCV) (m/sec) of common peroneal nerve (CPN) | 12 weeks
NCV (m/sec) of tibial nerve | 12 weeks
Distal latency (millisecond) of superficial peroneal nerve (SPN) | 12 weeks
Distal latency (millisecond) of sural nerve | 12 weeks
Sensory amplitude (microvolt) of SPN | 12 weeks
Sensory amplitude (microvolt) of sural nerve | 12 weeks
Motor amplitude (microvolt) of CPN | 12 weeks
Motor amplitude (microvolt) of tibial nerve | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mesbah Shams, M.D., Study Chair — Research Center for Traditional Medicine & History of Medicine - Shiraz University of Medical Sciences
Locations (2):
- Iran (2):
  - Department of Physical Medicine and Rehabilitation - Shiraz University of Medical Sciences, Shiraz, Fars
  - Research Center for Traditional Medicine and History of Medicine-Shiraz University of Medical Sciences, Shiraz, Fars